CLINICAL TRIAL: NCT04488562
Title: Home Monitoring and Evaluation After Admission for COVID-19 in the Netherlands
Acronym: HOMECOMIN'
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Leiden University Medical Center (Other); Amsterdam UMC, location VUmc (Other); Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2020-0318
Record Dates: First submitted 2020-06-02; First posted 2020-07-28 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Pulmonary Fibrosis
Keywords: Home monitoring
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19: Patients with proven COVID-19 and abnormalities on chest X-Ray/HRCT, admitted at the hospital. Patients are included around the time of discharge from the hospital or at their regular outpatient clinic visit 6 weeks after discharge, depending on the clinical status of the patient at time of discharge.

SUMMARY:
To date, little is known about the short and long-term complications of COVID-19. In order to obtain more insights in disease course and recovery of COVID-19 and to improve care after hospital admission, patients with COVID-19 will be monitored at home using an online home monitoring program for a period of 1 year.

DETAILED DESCRIPTION:
Patients with COVID-19 have a variable disease course and recovery. After the SARS coronavirus outbreak in 2003, many patients developed pulmonary fibrosis. Emerging data from the COVID-19 outbreak suggests that a substantial number of patient will likely develop pulmonary fibrosis. However, much is still unknown (e.g. the percentage of patients who develop pulmonary fibrosis, progression of fibrosis). Since we have little knowledge on the disease course and long-term complications of COVID-19, it is very important to properly monitor patients after hospital admission. An online home monitoring program could be an efficient way to monitor disease course of COVID-19 and provide insights in the long-term effects of COVID-19.

In this prospective, observational multi center study we aim to include 150 patients that were admitted in the hospital with abnormalities on chest X-ray/HRCT due to COVID-19. Based on their clinical status, patients will be either included at time of discharge from the hospital or at time of their regular outpatient clinic visit, 6 weeks after discharge from the hospital. Patients will be monitored for a period of 1 year after admission, after signing informed consent. Home monitoring, consisting of real-time lung function measures and PROMs, has been developed and validated for patients with pulmonary fibrosis; home monitoring was feasible, FVC measurements were reliable and patient satisfaction was high.

Patients are asked to fill in a diary once weekly (consisting of Visual Analogue Scales on cough, dyspnea, fatigue, general well-being, and temperature and oxygen measurements) and measure their lung function (FVC) at home every week with a home spirometer (Spirobank Smart, MIR, Italy) (duration + -2 min). The spirometer is connected via Bluetooth with the secured app and results can be sent directly to the study team. Patients are instructed to contact the hospital using a secured eConsult if they have worsening complaints and/or have a decrease in saturation or lung function.

Patients are asked to fill complete short validated questionnaires (ABC tool, EQ5D-5L, Fatigue Assessment Scale and Global rating of change, duration + - 10 minutes) in the app, at time of discharge, 6 weeks, 3 months, 6 months, 9 months and 12 months after discharge.

Demographic data, clinical characteristics, lung function results, radiology data and data about medication will be collected from the electronic patient file during regular outpatient clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital with proven COVID-19 infection
* Abnormalities on Chest X-ray/HRCT due to COVID-19 infection

Exclusion Criteria:

* Not able to speak, read or write in the native language of the country where the patient is included
* Not able to comply to the study protocol, according to the judgement of the investigator and/or patient
* No access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients admitted at the Erasmus Medical Center, Leiden University Medical Center and the Amsterdam University Medical Center, location VUMC, with proven COVID-19 infection and abnormalities on Chest X-ray/HRCT due to COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
VAS | 3 months
  Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
VAS | 6 months
  Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
VAS | 12 months
  Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
Temperature | 3 months
  Body temperature measured with an thermometer
Oxygen measurements | 3 months
  Oxygen saturation measured with an pulse oximeter
Oxygen measurements | 6 months
  Oxygen saturation measured with an pulse oximeter
Oxygen measurements | 12 months
  Oxygen saturation measured with an pulse oximeter
Forced Vital Capacity (FVC) home spirometry in % | 3 months
  FVC change measured with home spirometry at 3 months (in %)
Forced Vital Capacity (FVC) home spirometry in L | 3 months
  FVC change measured with home spirometry at 3 months (in L)
Forced Vital Capacity (FVC) home spirometry in % | 6 months
  FVC change measured with home spirometry at 6 months (in %)
Forced Vital Capacity (FVC) home spirometry in L | 6 months
  FVC change measured with home spirometry at 6 months (in L)
Forced Vital Capacity (FVC) home spirometry in L | 12 months
  FVC change measured with home spirometry at 12 months (in L)
Forced Vital Capacity (FVC) home spirometry in % | 12 months
  FVC change measured with home spirometry at 12 months (in %)
Forced Vital Capacity (FVC) hospital spirometry in % | 3 months
  FVC change measured with hospital spirometry and saturation at 3 months (in %)
Forced Vital Capacity (FVC) hospital spirometry in L | 3 months
  FVC change measured with hospital spirometry and saturation at 3 months (in L)
Forced Vital Capacity (FVC) hospital spirometry in % | 6 months
  FVC change measured with hospital spirometry and saturation at 6 months (in %)
Forced Vital Capacity (FVC) hospital spirometry in L | 6 months
  FVC change measured with hospital spirometry and saturation at 6 months (in L)
Forced Vital Capacity (FVC) hospital spirometry in % | 12 months
  FVC change measured with hospital spirometry and saturation at 12 months (in %)
Forced Vital Capacity (FVC) hospital spirometry in L | 12 months
  FVC change measured with hospital spirometry and saturation at 12 months (in L)
Adherence to weekly home spirometry | 1 year after inclusion
  The percentage of patients completed weekly home spirometry
EQ5D | Baseline
  The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status
EQ5D | 6 weeks
  The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status
EQ5D | 3 months
  The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status
EQ5D | 6 months
  The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status
EQ5D | 9 months
  The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status
EQ5D | 12 months
  The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status
FAS | Baseline
  Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
FAS | 6 weeks
  Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
FAS | 3 months weeks
  Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
FAS | 6 months weeks
  Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
FAS | 9 months weeks
  Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
FAS | 12 months weeks
  Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
GRoC | Baseline
  Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
GRoC | 6 weeks
  Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
GRoC | 3 months
  Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
GRoC | 6 months
  Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
GRoC | 9 months
  Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
GRoC | 12 months
  Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
ABC tool | Baseline
  Questionnaire consisting of five domains: symptoms, functional state, mental state, emotions and fatigue, smoking status, exacerbations, dyspnoea, body mass index, lung function and self-reported physical activity. Outcomes are visualized using coloured balloons. green balloons indicate a satisfactory score, red balloons a low score and orange balloons an intermediate score. Grey balloons represent the balloons of previous visits.
ABC tool | 6 weeks
  Questionnaire consisting of five domains: symptoms, functional state, mental state, emotions and fatigue, smoking status, exacerbations, dyspnoea, body mass index, lung function and self-reported physical activity. Outcomes are visualized using coloured balloons. green balloons indicate a satisfactory score, red balloons a low score and orange balloons an intermediate score. Grey balloons represent the balloons of previous visits.
ABC tool | 3 months
  Questionnaire consisting of five domains: symptoms, functional state, mental state, emotions and fatigue, smoking status, exacerbations, dyspnoea, body mass index, lung function and self-reported physical activity. Outcomes are visualized using coloured balloons. green balloons indicate a satisfactory score, red balloons a low score and orange balloons an intermediate score. Grey balloons represent the balloons of previous visits.
ABC tool | 6 months
  Questionnaire consisting of five domains: symptoms, functional state, mental state, emotions and fatigue, smoking status, exacerbations, dyspnoea, body mass index, lung function and self-reported physical activity. Outcomes are visualized using coloured balloons. green balloons indicate a satisfactory score, red balloons a low score and orange balloons an intermediate score. Grey balloons represent the balloons of previous visits.
ABC tool | 9 months
  Questionnaire consisting of five domains: symptoms, functional state, mental state, emotions and fatigue, smoking status, exacerbations, dyspnoea, body mass index, lung function and self-reported physical activity. Outcomes are visualized using coloured balloons. green balloons indicate a satisfactory score, red balloons a low score and orange balloons an intermediate score. Grey balloons represent the balloons of previous visits.
ABC tool | 12 months
  Questionnaire consisting of five domains: symptoms, functional state, mental state, emotions and fatigue, smoking status, exacerbations, dyspnoea, body mass index, lung function and self-reported physical activity. Outcomes are visualized using coloured balloons. green balloons indicate a satisfactory score, red balloons a low score and orange balloons an intermediate score. Grey balloons represent the balloons of previous visits.

SECONDARY OUTCOMES:
Correlation between FVC, HRCT patterns, symptoms and quality of life | 3 months
  Correlation between FVC, HRCT patterns, symptoms and quality of life
Correlation between FVC, HRCT patterns, symptoms and quality of life | 6 months
  Correlation between FVC, HRCT patterns, symptoms and quality of life
Correlation between FVC, HRCT patterns, symptoms and quality of life | 12 months
  Correlation between FVC, HRCT patterns, symptoms and quality of life
Predictors for the course of recovery of COVID-19 infection after hospital admission | 12 months
  Predictors for the course of recovery of COVID-19 infection after hospital admission
Satisfaction of patients and caregivers with the use of a home monitoring system | 12 months
  Healthcare provider and patient satisfaction and experience with the online application. Patients and healthcare providers are asked about their experiences and opinions on homemonitoring.

CONTACTS AND LOCATIONS:
Overall Officials: M.S. Wijsenbeek, dr, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Amsterdam University Center - location VUmc, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam